CLINICAL TRIAL: NCT07007325
Title: Prospective Feasibility Pilot Study Evaluating the Value of [68Ga]Ga-PENTIXAFOR PET-CT in Patients With Metastatic Small Cell Lung Cancer (SCLC) at Diagnosis and Disease Progression
Acronym: PASSIFLORE
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICO-2023-16
Record Dates: First submitted 2025-03-20; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Small Cell Lung Carcinoma (SCLC)
Keywords: Small Cell Lung Carcinoma (SCLC); [68Ga]Ga-PentixaFor; immunohistochemistry (IHC); CXCR4 expression; [18F]FDG; Safety
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-PentixaFor (Experimental): The patient receives a single dose I.V. injection of [68Ga]Ga-PentixaFor 150 (± 50) MBq, corresponding to a peptide mass dose of ≤ 50 μg per administration.
  Interventions: Drug: [68Ga]Ga-PentixaFor

INTERVENTIONS:
Drug: [68Ga]Ga-PentixaFor — [68Ga]Ga-PentixaFor PET-CT

SUMMARY:
[68Ga]Ga-PentixaFor PET-CT will be performed in patients with Small cell lung cancer (SCLC) to confirm the targeting of CXCR4 by [68Ga]Ga-PentixaFor

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) accounts for approximately 15% of lung cancers, but remains a cancer with a poor prognosis, often detected at a metastatic stage and associated with a high rate of early recurrence.

Therapeutic options for unresectable SCLC are limited and essentially rely on first-line radiochemotherapy for limited disease or chemo-immunotherapy, possibly supplemented by radiotherapy, for extensive disease.

CXCR4 is a chemokine receptor that is highly expressed in this cancer. By targeting CXCR4 with [177Lu]Lu-PentixaTher or [90Y]Y-PentixaTher, patients with SCLC could benefit from a new type of treatment in this indication: Peptide Receptor Radionuclide Therapy (PRRT).

However, there is a need for a preliminary diagnostic study due to a lack of published data.

[68Ga]Ga-PentixaFor is an experimental compound that binds with high affinity to CXCR4 and appears to be a promising candidate for PET-CT imaging of SCLC. This initial step is crucial to confirm CXCR4 targeting by [68Ga]Ga-PentixaFor before considering PRRT with therapeutic radionuclides such as Lu-177 or Y-90 in future trials.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed before performing any trial specific procedure.
2. Male or female, age ≥ 18 years at time of study entry.
3. Patient with histologically proven small cell lung carcinoma, inoperable, non-pre-treated.
4. Metastatic disease documented by conventional imaging and/or [18F]FDG PET-CT with at least one metastatic measurable lesion (RECIST 1.1). Patients eligible for 1st line metastatic treatment.
5. Availability of tissue material (primary lesion and/or metastatic site) to allow additional immunohistochemical studies.
6. PS < 2.
7. Consent to use a contraception method for at least 3 months after each administration of [68Ga]Ga-PentixaFor.
8. Adequate Organ function confirmed by laboratory test results allowing for safe the [68Ga]Ga-PentixaFor administration.
9. Life expectancy greater than 3 months.
10. Patient has valid health insurance.
11. Patient willing and able to comply with the protocol throughout the duration of the study, including during treatment and scheduled visits and examinations, including follow-up.

Exclusion Criteria:

1. History of cancer in the 3 years prior to entry into the trial other than basal cell carcinoma of the skin or carcinoma in situ of the cervix.
2. History of anti-cancer treatments such as chemotherapy, radiotherapy or immunotherapy as well as other clinical trials for SCLC before the first [68Ga]Ga-PentixaFor PET-CT imaging.
3. Inability to lie still for at least 1 hour, or known claustrophobia.
4. Serious non-malignant disease (e.g., psychiatric, infectious, autoimmune, or metabolic) which may interfere with study objectives or patient safety or compliance, in the judgment of the investigator.
5. Unstable diabetes with blood glucose > 2 g/L.
6. Known hypersensitivity to any active pharmaceutical agent or constituent of the [68Ga]Ga-PentixaFor and/or [18F]FDG product.
7. Body weight of less than 48 kg.
8. Mental impairment that may compromise the ability to give informed consent and comply with study requirements.
9. Pregnant, likely to be pregnant or breastfeeding woman.
10. Patient deprived of liberty, under judicial safeguard, under curatorship or placed under the authority of a guardian.
11. Disorder preventing understanding of trial information or informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the concordance of tumoral lesions detected between [68Ga]Ga-PentixaFor PET-CT and [18F]FDG PET-CT, considered as the reference, performed at diagnosis | 30 days
  The concordance between the two techniques ([18F]FDG PET-CT and [68Ga]Ga-PentixaFor PET-CT) will be assessed by lesion at diagnosis.
  Cohen's Kappa coefficient will be calculated and accompanied by the probability of finding the same lesion on [68Ga]Ga-PentixaFor PET-CT knowing that it was present on [18F]FDG PET-CT (which may be similar to a measurement of sensitivity).

SECONDARY OUTCOMES:
Evaluate the concordance of tumoral lesions detected between [68Ga]Ga-PentixaFor PET-CT and [18F]FDG PET-CT, considered as the reference, performed at disease progression. | 24 months
  The concordance between the two techniques ([18F]FDG PET-CT and [68Ga]Ga-PentixaFor PET-CT) will be assessed by lesion at disease progression.
  Cohen's Kappa coefficient will be calculated and accompanied by the probability of finding the same lesion on [68Ga]Ga-PentixaFor PET-CT knowing that it was present on [18F]FDG PET-CT (which may be similar to a measurement of sensitivity).
Evaluate the diagnostic performances of [68Ga]Ga-PentixaFor PET-CT compared to [18F]FDG PET-CT considered as the reference. | 24 months
  The diagnostic performances will be assessed using the Specificity, at diagnosis time on one hand, and at disease progression time on the other hand.
Evaluate the correlation between semi-quantitative data of [68Ga]Ga-PentixaFor PET-CT with CXCR4 expression on biopsies, assessed by immunohistochemistry (IHC). | 24 months
  The correlation between the standardized uptake values (SUV) of [68Ga]Ga-PentixaFor -positive lesions and the biological expression of CXCR4 will be described by Spearman's ρ, at diagnosis and at disease progression time if data are available.
Describe the lesions identified by [68Ga]Ga-PentixaFor PET-CT and by [18F]FDG PET-CT. | 24 months
  The qualitative analysis will focus on lesion description in each major organ (lung, lymph node, bone marrow, brain...). Quantitative analysis will focus on continuous parameters at the lesion level (SUV, MTV, TLG and tumour-to-background ratio, etc.). The detection rate of tumour lesions will be calculated. This analysis will be conducted for each radiotracer at diagnosis time on one hand, and at disease progression time on the other hand.
Compare the number of lesions detected by [18F]FDG PET-CT and those detected by [68Ga]Ga-PentixaFor PET-CT. | 24 months
  A comparison of all lesions number detected between the two radiotracers will be conducted at diagnosis time on one hand, and at disease progression time on the other hand.
Description of the evolution of [68Ga]Ga-PentixaFor PET-CT data obtained at diagnosis and at disease progression time at the patient level. | 24 months
  Description of [68Ga]Ga-PentixaFor PET-CT data between diagnosis and disease progression time at the patient level will focus on the evolution of SUV value for each patient.
Assess safety profile of [68Ga]Ga-PentixaFor. | 24 months
  The occurrence and the frequency of adverse events of [68Ga]Ga-PentixaFor will be assessed up to 48 hours after [68Ga]Ga-PentixaFor administration. The safety is assessed using the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Description of the evolution of [68Ga]Ga-PentixaFor PET-CT data obtained at diagnosis and at disease progression time at the patient level. | 24 months
  Description of [68Ga]Ga-PentixaFor PET-CT data between diagnosis and disease progression time at the patient level will focus on the evolution of Total Lesion Uptake (TLU) value for each patient. TLU will be calculated from the total tumour volume and the lesions SUVmean.
Evaluate the diagnostic performances of [68Ga]Ga-PentixaFor PET-CT compared to [18F]FDG PET-CT considered as the reference. | 24 months
  The diagnostic performances will be assessed using the Positive Predictive Value (PPV), at diagnosis time on one hand, and at disease progression time on the other hand.
Evaluate the diagnostic performances of [68Ga]Ga-PentixaFor PET-CT compared to [18F]FDG PET-CT considered as the reference. | 24 months
  The diagnostic performances will be assessed using the Negative Predictive Value (NPV), at diagnosis time on one hand, and at disease progression time on the other hand.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Institut de cancérologie de l'ouest, Angers
  - CHU d'Angers, Angers
  - Institut de cancérologie de l'ouest, Saint-Herblain